CLINICAL TRIAL: NCT01338987
Title: Multi-Institutional Prospective Pilot Study of Lupron to Enhance Lymphocyte Immune Reconstitution Following Allogeneic Bone Marrow Transplantation in Post-Pubertal Children and Adults With Molecular Imaging Evaluation
Brief Title: Pilot Study of Leuprolide to Improve Immune Function After Allogeneic Bone Marrow Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Christopher Kanakry, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110136; 11-C-0136
Record Dates: First submitted 2011-04-19; First posted 2011-04-20 (Estimated); Results first posted 2019-04-23 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Myelodysplastic Syndrome; Acute Lymphocytic Leukemia; Acute Myelogenous Leukemia; Chronic Myelogenous Leukemia; Chronic Myelomonocytic Leukemia
Keywords: FLT; Leuprolide; Thymic Renewal; Stem Cell Transplant; Acute Lymphocytic Leukemia; Acute Myelogenous Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myelomonocytic, Chronic | interventions — Leuprolide; alovudine; Cyclophosphamide; Methotrexate; Tacrolimus; Whole-Body Irradiation; Busulfan; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm1 First Transplt/males/leuprolide/+/-FLT Imaging (Active Comparator): Males randomized to leuprolide for first transplant.
  [18F]fluorothymidine (FLT) imaging
  Interventions: Procedure: First Allogeneic Bone Marrow Transplant (BMT); Drug: Leuprolide; Drug: 18F FLT; Drug: Cyclophosphamide; Drug: Methotrexate; Drug: Tacrolimus; Radiation: Total Body Irradiation
- Arm2 First Transplt/males/No Leuprolide/+/- FLT Imaging (Active Comparator): Males not receiving leuprolide for first transplant
  [18F]fluorothymidine (FLT) imaging
  Interventions: Procedure: First Allogeneic Bone Marrow Transplant (BMT); Drug: 18F FLT; Drug: Cyclophosphamide; Drug: Methotrexate; Drug: Tacrolimus; Radiation: Total Body Irradiation
- Arm3 First Transplt/females/leuprolide+/- FLT Imaging (Experimental): Females receiving leuprolide for first transplant.
  [18F]fluorothymidine (FLT) imaging
  Interventions: Procedure: First Allogeneic Bone Marrow Transplant (BMT); Drug: 18F FLT; Drug: Cyclophosphamide; Drug: Methotrexate; Drug: Tacrolimus; Radiation: Total Body Irradiation
- Arm4-Second Transplt/leuprolide and FLT Imaging (Experimental): Second transplant with leuprolide and [18F]fluorothymidine (FLT) imaging
  Interventions: Drug: Leuprolide; Drug: 18F FLT; Drug: Cyclophosphamide; Radiation: Total Body Irradiation; Drug: Busulfan; Drug: Fludarabine; Procedure: Second Allogeneic Bone Marrow Transplantation
- Healthy Volunteer - Arm 5 (No Intervention): Healthy Volunteer

INTERVENTIONS:
Procedure: First Allogeneic Bone Marrow Transplant (BMT) — First Allogeneic Bone Marrow Transplant
  Arms: Arm1 First Transplt/males/leuprolide/+/-FLT Imaging; Arm2 First Transplt/males/No Leuprolide/+/- FLT Imaging; Arm3 First Transplt/females/leuprolide+/- FLT Imaging
Drug: Leuprolide — Leuprolide: 30 mg intramuscular injection(for adult) or 11.25 mg (for patients <18 years) between day -13 and day -20 pre-bone marrow transplant but definitely prior to initiation of preparative regimen as a 4 month intramuscular injection for patients > 18 years and as a 3 month injection (adult preparation) for patients < 18 years
  Other Names: Lupron
  Arms: Arm1 First Transplt/males/leuprolide/+/-FLT Imaging; Arm4-Second Transplt/leuprolide and FLT Imaging
Drug: 18F FLT — For the first 23 patients undergoing 1st bone marrow transplant (BMT):[18F]fluorothymidine (18F FLT): 0.07 mCi/kg with a maximum of 3 mCi On day + 28 (+/- 5 days) For 2nd BMT: 18F FLT: 0.07 mCi/kg with a maximum of 3 mCi On day -1, + 28, day 60 and at relapse (+/- 5 days)
  Other Names: [18F]fluorothymidine
  Arms: Arm1 First Transplt/males/leuprolide/+/-FLT Imaging; Arm2 First Transplt/males/No Leuprolide/+/- FLT Imaging; Arm3 First Transplt/females/leuprolide+/- FLT Imaging; Arm4-Second Transplt/leuprolide and FLT Imaging
Drug: Cyclophosphamide — Cyclophosphamide: 60 mg/kg intravenous (IV) on days -4 and -3 (for Adults > 22 years) or Cyclophosphamide: cyclophosphamide 50 mg/kg IV, Days -5, -4, -3, -2. (For Pediatric </= 22 years)
  Other Names: Cytoxan
  Arms: Arm1 First Transplt/males/leuprolide/+/-FLT Imaging; Arm2 First Transplt/males/No Leuprolide/+/- FLT Imaging; Arm3 First Transplt/females/leuprolide+/- FLT Imaging; Arm4-Second Transplt/leuprolide and FLT Imaging
Drug: Methotrexate — Methotrexate:10 mg/m(2) intravenous (IV) on day +1, and 5 mg/m(2) IV Days + 3, 6, 11
  Other Names: Trexall
  Arms: Arm1 First Transplt/males/leuprolide/+/-FLT Imaging; Arm2 First Transplt/males/No Leuprolide/+/- FLT Imaging; Arm3 First Transplt/females/leuprolide+/- FLT Imaging
Drug: Tacrolimus — Tacrolimus:0.02 mg/kg/day continuous intravenous infusion (CIV) on day -1.
  Other Names: Prograf
  Arms: Arm1 First Transplt/males/leuprolide/+/-FLT Imaging; Arm2 First Transplt/males/No Leuprolide/+/- FLT Imaging; Arm3 First Transplt/females/leuprolide+/- FLT Imaging
Radiation: Total Body Irradiation — Total Body Irradiation (TBI) 1200 cGy fractionate twice daily (lung block) Days -8, -7, -6, -5 (adult), -9, -8, -7, -6 (ped)
  Arms: Arm1 First Transplt/males/leuprolide/+/-FLT Imaging; Arm2 First Transplt/males/No Leuprolide/+/- FLT Imaging; Arm3 First Transplt/females/leuprolide+/- FLT Imaging; Arm4-Second Transplt/leuprolide and FLT Imaging
Drug: Busulfan — Second choice is Busulfan (with goal steady state of 800-1000) with fludarabine or cyclophosphamide at myeloablative dosing or non-myeloablative dosing.
  Other Names: Busulfex
  Arms: Arm4-Second Transplt/leuprolide and FLT Imaging
Drug: Fludarabine — Given with Busulfan as alternative to cyclophosphamide in second transplant setting only
  Other Names: Fludara
  Arms: Arm4-Second Transplt/leuprolide and FLT Imaging
Procedure: Second Allogeneic Bone Marrow Transplantation — Second Allogeneic Bone Marrow Transplantation
  Arms: Arm4-Second Transplt/leuprolide and FLT Imaging

SUMMARY:
Background:

* One way to treat certain cancers of the blood and immune system is to give a patient stem cells from the bone marrow of a donor whose genes are very similar but not identical to the patients. One problem with these transplants is that the new immune cells may not work as well in the recipient as they did in the donor. The result may be that the immune system will not work as well. This can increase the risk of severe infections and other complications.
* Researchers are studying the use of drugs that lower hormone levels and may allow the immune system to recover in a way that improves white blood cell function. In this study they will be looking at the drug leuprolide, a drug that lowers estrogen or testosterone levels, to see if it might improve the function of the newly transplanted cells.

Objectives:

* To determine whether leuprolide improves immune system function after bone marrow transplant from a donor with similarities in their immune cells (matched to each other).
* To evaluate the effectiveness of a nuclear medicine test with a radiotracer drug 3-deoxy-3 18F-fluorothymidine (FLT) in imaging studies. FLT will be used to image the immune system function in patients who have received bone marrow from the donor.

Eligibility:

* People between 15 (or as young as 9 in those who have gone through puberty) and 55 years of age. These patients must have acute myelogenous leukemia, acute lymphocytic leukemia, high-risk myelodysplastic syndrome, chronic myelomonocytic leukemia, or chronic myeloid leukemia. They must also be eligible for a bone marrow transplant.
* Genetically similar donors for the patients who are eligible for a transplant.

Design:

* People taking part in the study will be screened with a physical examination, medical history, blood and urine tests, and imaging studies. Patients who are not in remission or who require a bone marrow donor search may receive chemotherapy first.
* Donors will provide bone marrow for transplant according to standard bone marrow transplant (BMT) procedures.
* All women and half of the men will receive regular leuprolide doses 2 weeks before BMT to suppress hormone function.
* All recipients will receive 4 days of radiation followed by 2-4 days of chemotherapy before the bone marrow transplant (depending on age). Recipients will also receive other drugs to prevent transplant rejection and other complications of transplantation.
* Recipients will be monitored in the hospital for 4 weeks after transplant with blood tests and other studies.
* Some recipients will have an imaging study with FLT during the protocol. These imaging studies will take place before the transplant, on days 5 and 28 after transplant, and at a later time to be determined by the study researchers.
* Following discharge, participants will be monitored closely for up to 6 months, with regular but less frequent followup visits for at least 5 years. Study-related medications, including vaccinations for the new immune system, will be provided by the National Institutes of Health during the hospital stay and after discharge.

DETAILED DESCRIPTION:
Background:

* Impaired lymphocyte immune reconstitution is associated with morbidity and mortality following allogeneic bone marrow transplant (BMT).
* Data suggest that one of the limitations of immunity after BMT is the lack of thymus recovery and proper B cell development.
* Androgen withdrawal has been shown to enhance T and B lymphopoiesis.
* Leuprolide is an approved, safe, gonadotropin releasing hormone (GnRH) agonist/antagonist.
* Noninvasive imaging modalities to study immune reconstitution would be invaluable to predict optimal or impaired immune recovery permitting early institution of therapies.
* FLT is 3-deoxy-3 18F-fluorothymidine, a radiolabeled thymidine analogue that illustrates dividing hematopoietic cells and may predict immune recovery after allogeneic BMT.
* FLT has been used safely in patients who have received intensive chemotherapy.

Objectives:

* Primary: To determine if leuprolide improves B lymphocyte reconstitution after first BMT.
* Primary: To assess whether 18F FLT positron emission tomography (PET)/computed tomography (CT) could predict early engraftment/immune reconstitution in marrow and thymus after allogeneic BMT.
* Primary: To assess safety of leuprolide after 2nd BMT evaluated in a separate arm.

Eligibility:

* Patients > 9 years old and pubertal and/or >15 year and less than or equal to 55 years, with aggressive leukemia (Acute Myelogenous Leukemia (AML), myelodysplastic syndromes (MDS) with high risk cytogenetics, Acute Lymphocytic Leukemia (ALL), CMML, certain CML) requiring BMT will be enrolled at National Cancer Institute (NCI).
* At University of Oklahoma, Age > 17 years old and less than or equal to 55 years for recipient.
* Patients > 4 and < 24 years with the above diseases will be enrolled at Children's National Medical Center (CNMC).

Design:

* This is a prospective pilot study, the primary aims of which are: 1) to assess whether leuprolide enhances lymphocyte recovery after first BMT, 2) whether FLT imaging can be used to predict engraftment/immune reconstitution after first transplant, and 3) whether leuprolide and FLT are tolerable for second HSCT.
* At NCI and Univ of Oklahoma, post-pubertal pediatric male patients (<18 years) will be randomized to receive a 3 month (11.25 mg) injection and adult male patients will be randomized to receive 4-month preparation of leuprolide (30 mg) or placebo two weeks before the preparative regimen for first BMT. Women and all individuals undergoing 2nd BMT will receive leuprolide at these doses per age and be evaluated in the treated cohort. At Children's National Medical Center, the patients will not receive leuprolide outside of the context of clinical care and will receive myeloablative BMT as per standard of care with FLT imaging for engraftment as the only primary endpoint.
* A target of 68 evaluable adult patients will be enrolled on this trial, which may necessitate up to 118 patients (118 donors) enrolled to reach this target at NCI and University of Oklahoma. A total of 10 pediatric patients will be enrolled at Children's National Medical Center for FLT imaging only. Sixteen patients will be enrolled to undergo second BMT.
* At NCI, adults greater than 18 years old both female and adult male patients undergoing 2nd BMT will receive 4-month preparation of leuprolide (30 mg) two weeks before the preparative regimen. All patients will undergo FLT imaging to evaluate whether this may predict BMT response or failure (relapse). This will be a pilot arm of 16 patients total.
* The planned length of this trial is 7 years with interim analyses at day 100 and day 365.
* Some of the patients are anticipated to be evaluated using FLT (to include only patients needed for the immunological primary endpoint, not increasing total patient numbers). 23 adult NCI patients in total will undergo FLT PET/CT imaging on day -1, at day +5 or day +9, at 4 weeks, and at a future point to include evidence of graft-versus-host disease (GVHD) relapse, or immune recovery. An estimated 50 patients (including subset of the 23 patients undergoing serial scanning) will be imaged approximately at 1 year for evaluation of thymus reconstitution. The total possible numbers will include no more than 118 patients to achieve the 68 evaluable adults for the immunological primary endpoint. However, all 23 FLT PET/CT imaged NCI patients will undergo a single 1 year FLT for evaluation of thymus reconstitution. Up to 10 pediatric patients at CNMC will undergo FLT PET/CT imaging on Day -1, day+9, and day +28 (if possible). Initial images will be correlated with engraftment and other secondary endpoints.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

INCLUSION CRITERIA: TRANSPLANT RECIPIENT

1. At National Institutes of Health (NIH). Age greater than or equal to 15 years old and/or greater than or equal to 9 years old and pubertal and less than or equal to 55 years for recipient. Pubertal is defined by: prior menses at any time (females), documentation of clinical Tanner stage greater than 2 at some point pre-chemotherapy or at the current visit. (At this point, sex steroids have been produced for a few years which have driven initial pubertal development). Tanner 2 is defined as: breast buds for females with coarse pubic hair, and coarse pubic hair and testes > 2.5cm for males.
2. At Children's National Medical Center only: age > 4 years old and < 24.
3. At University of Oklahoma: Age greater than or equal to 17 years old and less than or equal to 55 years for recipient.
4. A diagnosis of a hematologic malignancy for which stem cell transplant is standard of care:

4.1. Acute Lymphocytic Leukemia (ALL)

Adult: (greater than or equal to 22 years) greater than or equal to compete remission 2 (CR2) OR complete remission 1 (CR1) with:

* Matched sibling donor for recipient treated on adult leukemia regimen
* t(9:22) or bcr-abl+; t(4:11), t(1:19), t(8:14), 11q23 (MLL rearrangements) complex cytogenetics (5 or more chromosomal abnormalities), hypodiploidy (<44 chromosomes). Note that patients with ALL blast crisis who emerge from chronic myeloid leukemia (CML) are also eligible
* Primary induction failure, defined as failure to achieve CR with primary induction chemotherapy
* High white blood cell (WBC) (>30,000 for B-cell ALL and >100,000 for T-cell ALL) at diagnosis
* Persistence of minimal residual disease despite induction chemotherapy

Pediatric (< 22 years): greater than or equal to CR2 OR CR1 with high risk features

* Matched sibling donor for recipient treated on adult leukemia regimen
* Primary induction failure (M3 (>25% with greater 200 cells counted) marrow at day 29), M2 (5-25% blasts with greater than 200 cells counted) bone marrow or minimal residual disease (MRD) > 1% at day 29 who then fail at day 43 with either an M2 or M3 BM or MRD > 1%
* Persistent leukemia and t(9;22) (MRD >1% day 29 or MRD > 0.01% end consolidation)
* 11q23 (MLL) rearrangements detected by cytogenetic or polymerase chain reaction (PCR) at initial diagnosis who are slow early responders (M2/M3 at day 14 or MRD> 0.01% at day 29)
* Extreme hypodiploidy (< 44 chromosomes or deoxyribonucleic acid (DNA) index of <0.81) detected by cytogenetic/ploidy analysis

4.2 Acute Myelogenous Leukemia

Adult: (greater than or equal to 22 years) greater than or equal to CR2 OR CR1 with high one of the following risk features

-Adverse or intermediate-risk cytogenetics including:

1. Normal cytogenetics
2. complex karyotype (>2 abnormalities)
3. inv (3) or t (3;3); t(11;19)(q23;p13.1); +13; -17/17p-; -18; -20; (t(6;9); t(6;11); -7, 7q-; -5, 5q-; trisomy 8; t(3;5); t(9:11)(p22q23)
4. monosomy karyotype (presence of an autosomal monosomy in conjunction with at least one other autosomal monosomy or structural abnormality.
5. Any other karyotype EXCEPT t(8;21), t(9;11), inv(16), or t (16;16), and M3 (17; 17) unless ckit mutation present and then eligible.
6. AML emerging from CML (blast crisis) are eligible

   -Primary induction failure, defined as failure to achieve CR with primary induction chemotherapy
   * Secondary AML, defined as AML related to antecedent myelodysplastic syndrome (MDS), myeloproliferative neoplasms (MPN), or cytotoxic chemotherapy
   * Hyperleukocytosis (White blood cell (WBC) > 100,000 at diagnosis)
   * Mutations in the FMS-like tyrosine kinase 3 (FLT3) gene (FLT3-LM; FLT-ITDs)
   * Bilineage or biphenotypic leukemias are high risk features and eligible.

   Pediatric (< 22 years): greater than or equal to CR2 OR CR1 with a high risk feature including:

   -Primary induction failure (greater than or equal to 5% blasts in marrow after induction)
   * Persistent leukemia (>15% after first course of chemotherapy)
   * Complex karyotype, monosomy 7, or -5/-5q, FLT3 ITD-AR (>0.4) EXCEPT if also inv(16)/t(16;16), t(8,21)
   * Normal cytogenetics or abnormal cytogenetics EXCEPT if also inv(16)/t(16;16), t(8,21) are eligible for SIBLING transplant only
   * Bilineage or biphenotypic leukemias are high risk features and eligible.

   4.3. Myelodysplastic Syndrome Refractory Anemia with Excess Blasts (RAEB) 1 or 2; cytogenetics showing complex karyotype (3 or more abnormalities), monosomy 7/del(7q), or inv(3)/t(3q)/del(3q); or transfusion dependent.

   4.4. Chronic Myelomonocytic Leukemia

   4.5. Chronic Myelogenous Leukemia who have failed 2G- tyrosine kinase inhibitors (TKI)

   4.6. Standard pediatric indications for myeloablative transplantation for patients undergoing bone marrow transplant at Children's National Medical Center per institutional guidelines

   5. Disease status

   If patients are found to not be in remission at screening, then the patient may be returned to their primary hematologist/oncologist or may receive chemotherapy as per standard of care for the malignant disease. Patients for whom this would be their first allogeneic transplant must be in remission (< 5% malignant blasts in marrow and peripheral blood and no evidence of extramedullary disease) for transplant. Patients enrolled on this protocol for their second transplant do not need to have attained remission prior to transplant.

   6. Performance status: Karnofsky or Lansky performance status greater than or equal to 60% AND life expectance of greater than 3 months.

   7. Ability to give informed consent. For recipients and donors < 18 years of age, their legal guardian must give informed consent. Pediatric patients will be included in an age appropriate discussion in accordance with institutional guidelines.

   8 Hepatic function: Patients must have evidence of adequate liver function prior to enrollment defined by total bilirubin < 2.5 mg/dL (unless documented Gilbert's syndrome) AND transaminases less than or equal to 5 x the upper limit of normal for age appropriate indices.

   9. Renal function: Patients must have evidence of adequate renal function to proceed with stem cell transplant, creatinine clearance > 60 ml/min/1.73 m(2). Glomerular filtration rate (GFR) may also demonstrate adequate renal function.

   10. Left ventricular ejection fraction greater than or equal to 50% OR shortening fraction of greater than or equal to 27% demonstrated on 2-dimension (2D) echocardiogram or multi-gated acquisition scan (MUGA).

   11. Pulmonary function of Diffusing Capacity of the Lung for Carbon Monoxide (DLC0) adj/alveolar volume (VA) and forced expiratory volume 1 (FEV1) greater than or equal to 60% of normal indices for age and height unless the patient has a likely acute reversible etiology of decline and then DLCO adj/VA greater than or equal to 30% of normal. Pediatric patients unable to complete pulmonary function tests (PFTs) may be enrolled as per enrolling institution Standard Operating Procedure (SOP) for recipient guidelines.

   12. Patients with prior autologous stem cell transplants will be included. Patients with prior allogeneic stem cell transplants will be eligible for 2nd BMT if not previously transplanted with FLT on this study.

   13. Prior experimental systemic therapies must have been completed greater than 2 weeks prior to study entry.

   EXCLUSION CRITERIA: TRANSPLANT RECIPIENT
   1. History of psychiatric disorder which may compromise compliance with transplant protocol, or which does not allow for appropriate informed consent.
   2. Active infections not responding to therapy. All efforts should be made to clear the infection prior to enrollment.
   3. Clinically significant systemic illness with manifestations of significant organ dysfunction which in the judgment principal investigator (PI) or associate investigator (AI) would render the patient unlikely to tolerate the protocol therapy or complete the study.
   4. Presence of active malignancy from an organ system other than hematopoietic.
   5. Human immunodeficiency virus (HIV) infection.
   6. Chronic active hepatitis B infection. Patients may be hepatitis B core antibody positive but must be surface antigen negative and without active evidence of disease.
   7. Pregnant or lactating females will be excluded from this trial due to unknown risks to the developing fetus. Patients of child-bearing potential must use an effective form of contraception while on study.
   8. Sexually active individuals capable of becoming pregnant who are unable or unwilling to use effective form(s) of contraception during time enrolled on study and for 1 year post-transplant.
   9. History of prior Leuprolide intolerance. Note: patients ARE eligible if prior or current leuprolide exposure.

   INCLUSION CRITERIA: MATCHED RELATED TRANSPLANT DONOR
   1. Age greater than or equal to 2 and less than or equal to 60 years old and able to give consent or assent. For donors < 18 years old, the legal guardian must be able to provide informed consent and an evaluation by a Licensed Social Worker (LSW) or psychiatric personnel will be needed to determine willingness to participate. Pediatric patients will be included in an age appropriate discussion in accordance with institutional guidelines.
   2. Human leukocyte antigen (HLA)-matched related donor, excluding identical twins. Donors must be matched at least 7 loci out of 8 at the allele or antigen level excluding antigen DRB1 mismatch.
   3. Donor selection will be in accordance with National Institutes of Health (NIH)/Clinical Center (CC) Department of Transfusion Medicine criteria and must be able to medically endure stem cell collection or as per local institutional guidelines.
   4. Donors must be HIV negative, human T-cell leukemia-lymphoma virus (HTLV) negative, hepatitis B surface antigen (HBsA) negative.
   5. Donors must be physically able to and willing to tolerate marrow harvest collection preferably, or in the absence of this option, able and willing to donate via peripheral blood pheresis.

   EXCLUSION CRITERIA: MATCHED RELATED TRANSPLANT DONOR
   1. History of medical illness that in the estimation of the PI or Department of Transfusion Medicine (DTM) physician precludes donation of marrow.
   2. Anemia (Hemoglobin (Hb) < 10 gm/dl) or thrombocytopenia (< 100,000/ ul).
   3. Pregnant females (due to risk to fetus).
   4. Current psychiatric diagnosis that would compromise compliance with transplant protocol or precludes appropriate informed consent.
   5. Presence of any blood transmissible infectious disease that cannot be cleared prior to stem cell collection and poses an unacceptable risk for the recipient (excludes cytomegalovirus (CMV)).
   6. Active malignancy will exclude the donor. Any malignancy less than five years postremission will exclude the donor. Non-hematologic malignancies greater than 5 years ago will not exclude the donor. Any history of hematologic malignancy will be considered on a case by case basis.
   7. Any medical contraindication to anesthesia or marrow donation will exclude the donor.
   8. Donors receiving experimental therapy or investigational agents.
   9. Active autoimmune disease that in the opinion of the PI or AI would compromise the success of the transplant.

   INCLUSION CRITERIA- MATCHED UNRELATED DONOR
   1. Unrelated donor matched at HLA-A, B, C, and DR loci by high resolution typing (at 8/8 or 7/8 antigen/allele match) are acceptable donors.
   2. The evaluation of donors shall be in accordance with existing National Marrow Donor Program (NMDP) Standard Policies and Procedures at all institutions.

   INCLUSION CRITERIA- (18F) FLT CANDIDATE TRANSPLANT RECIPIENT
   1. Meets criteria for Transplant Recipient
   2. Age greater than or equal to 18 years old at National Cancer Institute (NCI), and age > 4 years and < 24 years at Children's National Medical Center
   3. Donor who is willing to undergo bone marrow or stem cell harvest.

   EXCLUSION CRITERIA- (18F) FLT CANDIDATE TRANSPLANT RECIPIENT

   1. History of prior fluorothymidine allergy or intolerance.

Ages: 4 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2011-04-19 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2020-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher G Kanakry, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (3):
- United States (3):
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - University of Oklahoma, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hakim FT, Cepeda R, Kaimei S, Mackall CL, McAtee N, Zujewski J, Cowan K, Gress RE. Constraints on CD4 recovery postchemotherapy in adults: thymic insufficiency and apoptotic decline of expanded peripheral CD4 cells. Blood. 1997 Nov 1;90(9):3789-98. PMID 9345067
- [Background] Hazenberg MD, Otto SA, de Pauw ES, Roelofs H, Fibbe WE, Hamann D, Miedema F. T-cell receptor excision circle and T-cell dynamics after allogeneic stem cell transplantation are related to clinical events. Blood. 2002 May 1;99(9):3449-53. doi: 10.1182/blood.v99.9.3449. PMID 11964316
- [Background] Storek J, Gooley T, Witherspoon RP, Sullivan KM, Storb R. Infectious morbidity in long-term survivors of allogeneic marrow transplantation is associated with low CD4 T cell counts. Am J Hematol. 1997 Feb;54(2):131-8. doi: 10.1002/(sici)1096-8652(199702)54:23.0.co;2-y. PMID 9034287
- [Result] Williams KM, Holter-Chakrabarty J, Lindenberg L, Duong Q, Vesely SK, Nguyen CT, Havlicek JP, Kurdziel K, Gea-Banacloche J, Lin FI, Avila DN, Selby G, Kanakry CG, Li S, Scordino T, Adler S, Bollard CM, Choyke P, Gress RE. Imaging of subclinical haemopoiesis after stem-cell transplantation in patients with haematological malignancies: a prospective pilot study. Lancet Haematol. 2018 Jan;5(1):e44-e52. doi: 10.1016/S2352-3026(17)30215-6. Epub 2017 Dec 14. PMID 29248669
- [Derived] Holter-Chakrabarty J, McNally L, Levine J, Ferrara J, Vesely SK, Kanakry CG, Garwe T, Han Z, Pandey M, Glover J, Wen Y, Gress R, Williams KM. 18F-FLT PET and Blood-based Biomarkers for Identifying Gastrointestinal Graft versus Host Disease after Allogeneic Cell Transplantation. Radiol Imaging Cancer. 2025 Jan;7(1):e240096. doi: 10.1148/rycan.240096. PMID 39670843
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-C-0136.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Males That Did Not Receive Leuprolide for 1st Transplant: Males undergoing first transplant who did not receive leuprolide.
- Males Randomized to Receive Leuprolide for 1st Transplant: Males undergoing first transplant who were randomized to receive leuprolide.
- Females That Received Leuprolide for 1st Transplant: Females undergoing first transplant who all received leuprolide.
- Matched Related Donors for Transplant: Individuals related to patients and who gave hematopoietic stem cells for patients receiving allogeneic bone marrow transplant on this study.
- Recipients of 2nd Transplant: Patients receiving second allogeneic bone marrow transplant on this study.
Period: Overall Study
Arm/Group | Males That Did Not Receive Leuprolide for 1st Transplant | Males Randomized to Receive Leuprolide for 1st Transplant | Females That Received Leuprolide for 1st Transplant | Matched Related Donors for Transplant | Recipients of 2nd Transplant
Started | 12 | 9 | 22 | 31 | 2
Completed | 10 | 8 | 20 | 31 | 2
Not Completed | 2 | 1 | 2 | 0 | 0
Not completed — enrolled on new protocol | 0 | 0 | 1 | 0 | 0
Not completed — Disease progression on study | 2 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Males That Did Not Receive Leuprolide for 1st Transplant | Males Randomized to Receive Leuprolide for 1st Transplant | Females That Received Leuprolide for 1st Transplant | Matched Related Donors for Transplant | Recipients of 2nd Transplant | Total
Number analyzed (Participants) | 12 | 9 | 22 | 31 | 2 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 0 | 3 | 0 | 4
  Between 18 and 65 years | 11 | 9 | 22 | 28 | 2 | 72
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (9.30) | 26.77 (5.71) | 36.05 (6.10) | 33.86 (11.49) | 23.05 (3.61) | 33.61 (10.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 22 | 17 | 0 | 39
  Male | 12 | 9 | 0 | 14 | 2 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 6 | 15 | 26 | 1 | 56
  Not Hispanic or Latino | 4 | 3 | 7 | 5 | 1 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1 | 0 | 2
  Asian | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 3 | 2 | 0 | 8
  White | 9 | 5 | 15 | 28 | 2 | 59
  More than one race | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 2 | 3 | 0 | 0 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 9 | 22 | 31 | 2 | 76

OUTCOME MEASURES:

1. Primary Outcome: Percentage of B Cells at One Year Post-transplant in Participants Who Did/Did Not Receive Leuprolide Following Bone Marrow Transplant (BMT)
Description: B cell percentage is defined as the percentage of lymphocytes that are B cells.
Time Frame: after first Bone Marrow Transplant, approximately 12 months post-transplant
Population: Only first BMT patients (SG1-3) with >1 year of follow-up without relapse were evaluable. Of evaluable patients, 5 males and 9 females received and 7 males did not receive Lupron. Reasons for patients being inevaluable were missing data (2) or insufficient follow-up due to death without relapse (3), relapse (11), or withdrawal (1) before 1 year.
Measure: Median (Full Range); unit: percentage of cells
Groups:
- Transplant Recipient: Patients receiving first allogeneic bone marrow transplant on this study.
Arm/Group | Transplant Recipient
Number analyzed (Participants) | 21
percentage of cells
  Males that received leuprolide: number analyzed (Participants) | 5
  Males that received leuprolide | 22.1 [2.2 to 30.7]
  Males that did not receive leuprolide: number analyzed (Participants) | 7
  Males that did not receive leuprolide | 21.9 [0.2 to 32.5]
  Females who all received leuprolide: number analyzed (Participants) | 9
  Females who all received leuprolide | 14.3 [2.1 to 50.5]

2. Primary Outcome: Time to Engraftment in First Transplant Recipients Only With Median Thoracic Spine Standardized Uptake Values (SUV) of 1.4 or Greater Than Those Patients With SUV's Less Than 1.4
Description: 18F-FLT imaging was performed serially on patients post transplant to identify the level of uptake of 18F-FLT at a day +5 to +12 scan and the day at which neutrophils recover to >500 (i.e., subclinical bone-marrow recovery within 5 days of Bone Marrow Transplantation (BMT infusion)). On each image for each patient, the region of interest was drawn within each thoracic medullary space (n=12), generating the SUV for each space. The mean of these was calculated for each scan. The analysis was the median of the means of the SUV of the thorax values of the day 5-12 scan (averaged the SUV of the thorax for each patient and then took the medians of these).
Time Frame: 18F FLT scan done between days +5 to +12 and then time from that scan to engraftment measured
Population: The pre-specified cohort for this endpoint was 23 first BMT recipients. Only 20 of 23 were evaluable due to inability to obtain the early scan (1) or early relapse (2). As pre-specified in the protocol, all 20 patients were analyzed together as the intention was to look at the imaging modality itself and not any effect of leuprolide.
Measure: Median (Full Range); unit: Days
Arm/Group | Transplant Recipient
Number analyzed (Participants) | 20
Days
  Patients with SUV 1.4 or greater: number analyzed (Participants) | 5
  Patients with SUV 1.4 or greater | 5 [3 to 13]
  Patients with SUV less than 1.4: number analyzed (Participants) | 15
  Patients with SUV less than 1.4 | 15 [8 to 22]
Statistical Analysis 1: Comparison: Transplant Recipient; Test type: Other; p = 0.0075, Wilcoxon's rank sum test

3. Primary Outcome: Number of Adverse Events Related to Study Drug Experienced by Participants After Second Bone Marrow Transplant (BMT)
Description: Serious and non-serious adverse events were assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: 12 months after second BMT
Population: Only the patients in the SG4 group who had a 2nd BMT had a primary endpoint of toxicity requiring leuprolide AE reporting.
Measure: Number; unit: Adverse Events
Groups:
- Transplant Recipient - 2nd Bone Marrow Transplant: Patients receiving second allogeneic bone marrow transplant on this study.
Arm/Group | Transplant Recipient - 2nd Bone Marrow Transplant
Number analyzed (Participants) | 2
Adverse Events | 0

4. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 79 months and 11 days.
Population: 40/45 transplant recipients and all 31 donors were evaluable for adverse events as five patients did not proceed to transplant after enrollment due to progression of disease in four cases and enrollment on a new protocol in one case.
Measure: Count of Participants; unit: Participants
Arm/Group | Males That Did Not Receive Leuprolide for 1st Transplant | Males Randomized to Receive Leuprolide for 1st Transplant | Females That Received Leuprolide for 1st Transplant | Matched Related Donors for Transplant | Recipients of 2nd Transplant
Number analyzed (Participants) | 10 | 8 | 20 | 31 | 2
Participants | 10 | 8 | 20 | 4 | 2

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 79 months and 11 days.
Description: 40/45 participants were evaluable for adverse events.
Arm/Group | Males That Did Not Receive Leuprolide for 1st Transplant | Males Randomized to Receive Leuprolide for 1st Transplant | Females That Received Leuprolide for 1st Transplant | Matched Related Donors for Transplant | Recipients of 2nd Transplant
All-Cause Mortality (participants affected / at risk) | 4/10 | 3/8 | 8/20 | 0/31 | 2/2
Serious Adverse Events (participants affected / at risk) | 5/10 | 6/8 | 15/20 | 2/31 | 2/2
Other Adverse Events (participants affected / at risk) | 10/10 | 8/8 | 20/20 | 4/31 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Males That Did Not Receive Leuprolide for 1st Transplant (N=10) | Males Randomized to Receive Leuprolide for 1st Transplant (N=8) | Females That Received Leuprolide for 1st Transplant (N=20) | Matched Related Donors for Transplant (N=31) | Recipients of 2nd Transplant (N=2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Corneal ulcer (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death NOS (General disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 5 (8) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Infections and infestations - Other, E.coli (blood, lungs) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Fever, neutropenia (Infections and infestations) | 1 (1) | 0 (0) | 5 (8) | 0 (0) | 0 (0)
Infections and infestations - Other, Influenza H1N1 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, Kaposi's sarcoma (HHV8) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, PCP Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, Parainfluenza III (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Presumed fungal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Pseudomonas bacter (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, RSV (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Stenotrophom maltophilia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Stenotrophomonas bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, adeno viremia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, presumed bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Candida glabrata in blood (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Lung infection (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other, acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal hemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 4 (6) | 0 (0) | 2 (3)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and Infestations - Other, Candida glabrata in blood (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Males That Did Not Receive Leuprolide for 1st Transplant (N=10) | Males Randomized to Receive Leuprolide for 1st Transplant (N=8) | Females That Received Leuprolide for 1st Transplant (N=20) | Matched Related Donors for Transplant (N=31) | Recipients of 2nd Transplant (N=2)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 2 (3) | 6 (8) | 0 (0) | 1 (2)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2) | 4 (4) | 6 (10) | 0 (0) | 1 (3)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 6 (24) | 4 (8) | 14 (45) | 0 (0) | 1 (3)
Alkaline phosphatase increased (Investigations) | 3 (3) | 1 (6) | 5 (6) | 0 (0) | 1 (1)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 9 (28) | 5 (28) | 12 (39) | 3 (3) | 2 (4)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 5 (14) | 3 (5) | 13 (36) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 3 (4) | 2 (2) | 5 (10) | 0 (0) | 1 (2)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
CPK increased (Investigations) | 1 (2) | 2 (3) | 1 (2) | 0 (0) | 0 (0)
Carbon monoxide diffusing capacity decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colonic ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Corneal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 1 (2) | 2 (2) | 5 (7) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 2 (4) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (5) | 5 (6) | 10 (12) | 0 (0) | 2 (3)
Dry eye (Eye disorders) | 1 (1) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endocrine disorders - Other, Hypoganadism (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 2 (3) | 7 (7) | 0 (0) | 1 (2)
Fever (General disorders) | 4 (5) | 2 (5) | 6 (7) | 0 (0) | 1 (1)
Fibrinogen decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, Melanotic Stool (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hallucinations (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hepatobiliary disorders - Other, Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary disorders - Other, Ductal injury consistent w/GVHD, portal hypertension (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatobiliary disorders - Other, acute liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatobiliary disorders - Other, liver GVHD (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (12) | 1 (1) | 5 (8) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (4) | 0 (0) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (4) | 1 (1) | 8 (9) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (3) | 1 (4) | 8 (9) | 0 (0) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 4 (5) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 6 (17) | 3 (5) | 10 (13) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 4 (5) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 8 (15) | 4 (6) | 12 (21) | 0 (0) | 2 (3)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, 6/24 Aeromonas infection of stool (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, Adenoviremia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Ascaris lubricoides in stool (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, BK cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, BK virus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Blood cultures were positive for GPC/bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Blood cx: CMV+ ; CMV reactivation (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, C. diff (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, C. diff PCR+ 4/21 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, C. diff PCR+ 6/5 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, CMV (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, CMV (blood) (Infections and infestations) | 2 (2) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Infections and infestations - Other, CMV (blood, BAL, GI) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, CMV colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Infections and infestations - Other, CMV reactivation (Infections and infestations) | 2 (2) | 0 (0) | 6 (6) | 0 (0) | 0 (0)
Infections and infestations - Other, CMV reactivation (1600 copies) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, CMV reactivation (blood) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, CMV reactivation +6350 copies (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, CMV reactivation and presumed CMV infection of GI. (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, CMV viremia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, CMV viremia, CMV gastritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, CMV-esophagitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Coagulase-negative Staph, Rhinovirus/enterovirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, Coronavirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, Coronavirus 229E (nasal wash, upper respiratory) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, E.coli (UTI) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, EBV+PCR 3600 copies (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, ESBL Klebsiella urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, ESBL bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Enteroaggregative E.coli (stool) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Enterococcus in blood (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, Enteropathogenic E.coli (stool) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, GI tract (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Geotricum Capitatum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Giardia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, HHV6 (CSF) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, HSV oral ulcers (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Human metapneumovirus (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Infections and infestations - Other, Hypotension (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Influenza B (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, Klebsiela pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Klebsiella, serratia, stenotrophomonas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, Lymphadenitis (inguinal lymph node) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, Mumps (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, NP wash - rhinovirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Nocardia pulmonary infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, PICC, S.mitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Pleseimonas shigelloides (stool) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Presumed fungal - BAL (pulmonary) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Pseudomonas aeruginosa (skin lesion) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, RSV (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, Rhino/enterovirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, Rhinovirus/enterovirus (NP wash) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Rotavirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, Rothia (Stomatococcus) mucilaginosus; (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — 1/2 bottles with GPC in pairs & chains
Infections and infestations - Other, STAPH EPI from CSF (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, Shiga-like E.coli (SREC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Staph epi, Enterococcus faecalis in blood (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Staph. Capitis product infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, THRUSH (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, VRE bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, VZV (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, VZV zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, Vancomycin-resistant Enterococcus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Varicella zoster (back, abdomen) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Varicella zoster- L thoracic area (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, adenovirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, adenovirus viremia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, bacterial vaginosis and C.albicans (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, bronchscopy - aspergillus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, clostridium tertium (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, coronaviral URI (intermittent) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, fungal (yeast in blood) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, lung microbiology (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, norovirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, pneumonia-unknown organism (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, presumed BK virus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, presumed bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, presumed fungal pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Infections and infestations - Other, presumed pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, presumed pneumonia, yeast infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, presumed viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, rhinovirus/enterovirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, staph aureus (sinusitis) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Clostridium difficile - stool (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Infections and infestations - Other, HHV-6 (alveolar inf.) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, Human rhinovirus/enterovirus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, Staph epidermitis in blood (port inf.) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, intermittent bacteremia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 5 (7) | 3 (4) | 5 (7) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Pain, bilateral shins/ankles R>L (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (6) | 1 (2) | 9 (13) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 10 (49) | 7 (32) | 15 (83) | 0 (0) | 2 (2)
Oral pain (Gastrointestinal disorders) | 3 (3) | 1 (3) | 4 (6) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Otitis externa (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 4 (5) | 2 (2) | 5 (5) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 10 (43) | 7 (53) | 14 (49) | 0 (0) | 2 (6)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychiatric disorders - Other, acute mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (5) | 3 (3) | 5 (5) | 0 (0) | 1 (1)
Rectal mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, renal insufficiency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Reproductive system and breast disorders - Other, Dyspareunia, Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Reproductive system and breast disorders - Other, Vaginal bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Reproductive system and breast disorders - Other, vaginal scarring and stenosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Serum amylase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 1 (2) | 3 (3) | 0 (0) | 1 (2)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Porokeratosis - buttocks (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, cGVHD, scleroderma, rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, pimple-llike lesions neck, fase, chest (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomal ulcer (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0)
Vascular disorders - Other, Anasarca B/L (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vascular disorders - Other, TAM-transfusion associated microangiopathy (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (5) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Weight gain (Investigations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (2) | 2 (5) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 10 (33) | 4 (46) | 16 (56) | 0 (0) | 2 (6)
Renal and urinary disorders - Other, membranous nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, pneumonia, presumed fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, BK virus (urine infection) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, CMV (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, staph aureus (sinusitis) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, E. coli (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2017-12-28): https://cdn.clinicaltrials.gov/large-docs/87/NCT01338987/Prot_SAP_000.pdf
  • Informed Consent Form: Donor consent (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/87/NCT01338987/ICF_003.pdf
  • Informed Consent Form: Recipient consent (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/87/NCT01338987/ICF_004.pdf